CLINICAL TRIAL: NCT02009397
Title: A Phase I/II Open-Label Study of Ipilimumab and GM-CSF Administered to Unresectable Stage IIIC and Stage IV Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Jason Chesney, Director, James Graham Brown Cancer Center, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-MEL-11-02 (Ipi2)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab and GM-CSF (Experimental): IV ipilimumab followed by subcutaneous GM-CSF, for up to 4 cycles
  Interventions: Drug: Ipilimumab; Drug: GM-CSF

INTERVENTIONS:
Drug: Ipilimumab
Drug: GM-CSF

SUMMARY:
The purpose of this study is to test the combination of Ipilimumab and GM-CSF. Both ipilimumab and GM-CSF are intended to work with the body's own immune system to attack melanoma cells in the body. This study will also demostrate how safe the combined drugs are when used to treat patients with Stage 3 or Stage 4 melanoma (metastatic melanoma), which cannot be removed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be entered in the study only if they meet all of the following criteria.

  1. Male or female patients ≥18 years of age;
  2. Patients with histological confirmed melanoma (Stage IIIC or Stage IV, American Joint Commission on Cancer);
  3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2;
  4. Life expectancy ≥3 months;
  5. At least 1 site of radiographically measurable disease by immune-related response criteria (irRC);
  6. Adequate hematologic, renal, and liver function as defined by laboratory values performed within 42 days prior to initiation of dosing:

     * Absolute neutrophil count (ANC) ≥1.0 x 109/L;
     * Platelet count ≥50 x 109/L;
     * Hemoglobin ≥8 g/dL;
     * Serum creatinine ≤3 x upper limit of normal (ULN)
     * Total serum bilirubin ≤2 x ULN;
     * Serum aspartate transaminase (AST/SGOT) or serum alanine transaminase (ALT/SGPT) ≤2x ULN, and ≤3 x ULN if liver metastases are present.
  7. Fertile males should use an effective method of contraception during treatment and for at least 3 months after completion of treatment, as directed by their physician;
  8. Pre-menopausal females and females <2 years after the onset of menopause should have a negative pregnancy test at Screening. Pre-menopausal females must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 90 days after the last dose of study drug. Females of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year;
  9. Before study entry, written informed consent must be obtained from the patient prior to performing any study-related procedures.

Exclusion Criteria:

* Patients will not be entered in the study for any of the following:

  1. Treatment with Denileukin Diftitox within 42 days prior to the start of Ipilimumab;
  2. Prior treatment with Ipilimumab;
  3. Known hypersensitivity to Ipilimumab or any of its components
  4. Received radiotherapy for non CNS disease within the 2 weeks prior to commencing study treatment or have not recovered from side effects of all radiation-related toxicities to Grade ≤1, except for alopecia;
  5. Steroids within one week prior to initiation of Ipilimumab.
  6. Pre-existing autoimmune colitis.
  7. Patients with an allograft requiring immunosuppression;
  8. Known positive human immunodeficiency virus (HIV)
  9. Pregnant, breast-feeding, or refusing double barrier contraception, oral contraceptives, or avoidance of pregnancy measures;
  10. Have any other uncontrolled infection or medical condition that could interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chesney, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipilimumab and GM-CSF: IV ipilimumab followed by subcutaneous GM-CSF, for up to 4 cycles
  Ipilimumab
  GM-CSF
Period: Overall Study
Arm/Group | Ipilimumab and GM-CSF
Started | 26
Completed | 6
Not Completed | 20
Not completed — Protocol Violation | 6
Not completed — Death | 8
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab and GM-CSF
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 58 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Immune-related Overall Response Rate (irORR)
Time Frame: assessed at baseline and at 4 weeks (±1 week) following the last administration of Ipilimumab
Measure: Number; unit: participants
Arm/Group | Ipilimumab and GM-CSF
Number analyzed (Participants) | 20
participants | 20

ADVERSE EVENTS:
Arm/Group | Ipilimumab and GM-CSF
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes